CLINICAL TRIAL: NCT01628055
Title: IVIG in Acute Ischemic Stroke: A Pilot Study
Acronym: IVIG/AIS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: difficult recruitment and new black box warning for IVIG
Sponsor: Inova Health Care Services (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVIG/AIS-IFH-MB-CSL
Record Dates: First submitted 2012-06-14; First posted 2012-06-26 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Stroke
Keywords: IVIg; Acute Ischemic Stroke; Stroke; CVA; Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Immunoglobulins, Intravenous; gamma-Globulins; Fluid Therapy; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Privigen (Experimental): The IVIG preparation to be used is 10% liquid (Privigen). IVIG will be applied at a dose of 1.0g/kg, which is approximately 1/2 of the optimal dose used for other immuno/inflammatory indications. The infusion will start at 0.5 ml/kg/hr for the first 30 minutes, to watch for the signs of hypersensitivity to immunoglobulins, and then increased to 2.5 ml/kg/hr, two times slower than the recommended rate indicated in the product package insert (5 ml/kg/hr). Such a low, single dose has not been associated with hyperviscosity and together with a slow infusion will safeguard against occurrence of adverse events related to IVIG infusions. They will receive a total of 1g/kg and depending on patient's weight, it will take between 3.5 to 4+ hours to infuse that amount.
  Interventions: Biological: Privigen
- Normal Saline (Placebo Comparator): The placebo is the normal saline. Since saline solution will be infused at the volume equivalent to that in which the intended dose of immunoglobulin molecules will be delivered, the placebo (comparator) arm will also serve as a control for the volume of fluid infused to the treatment arm participants.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Privigen — 10% liquid intravenous immunoglobulin at a single dose of 1.0g/kg, run at 0.5ml/kg/hr for the first 30 minutes, then increased to 2.5ml/kg/hr until complete (~3-4 hours depending on weight).
  Other Names: IVIg; Immune Globulin Intravenous (Human); Immune Globulin Intravenous (Human), 10% Liquid
  Arms: Privigen
Other: Normal Saline — Normal Saline is a sterile, nonpyrogenic solution for fluid and electrolyte replenishment. It contains no antimicrobial agents. The pH is 5.0 (4.5 to 7.0).
  It contains 9 g/L Sodium Chloride with an osmolarity of 308 mOsmol/L and 154 mEq/L Sodium and Chloride.
  The infusion will start at 0.5 ml/kg/hr for the first 30 minutes and then increased to 2.5 ml/kg/hr for 3-4 hours.
  Other Names: 0.9% Sodium Chloride Solution
  Arms: Normal Saline

SUMMARY:
The purpose of the study is to evaluate the ability of IVIG to affect the rate of progression of brain ischemia, as evidenced by neuroimaging.

The results of an ongoing epidemiological study indicate that patients with primary immunodeficiency (PID) on IVIG replacement therapy have an overall prevalence of stroke that is 5 times less than in the general population. Even more striking is the absence of stroke in IVIG-treated PID patients over 65, while in the same general population age group the stroke prevalence goes up to 8.1%. This suggests that the degree of stroke protection correlates with the length of IVIG treatment, since older PID patients have been treated with IVIG significantly longer than younger ones.

DETAILED DESCRIPTION:
Two pre-clinical studies demonstrated the effectiveness of IVIG preparations in improving the clinical outcome of stroke and at the same time provided evidence of the role of complement fragments in the pathogenesis of ischemia-induced brain damage. Scavenging of these active fragments by IVIG is the likely mechanism of beneficial effect. In one of these studies CSL's own Privigen preparation was used. Considering that it exhibited in-vitro scavenging abilities more pronounced than several other IVIG preparations, and that its in-vivo scavenging capacity was also proven in a relevant animal model, a need to test this preparation in stroke patients is warranted. In addition, activation of complement and the level of activated fragments in humans seem to correlate with the severity of the disease, making them an ideal therapeutic target.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of neurological symptoms between 4.5 and 8 hours
2. Male or Female age 45 -75 years old
3. Score of 10-15 points on the National Institutes of Health Stroke Scale (NIHSS) with clinical signs suggestive of ischemic stroke
4. Acute brain ischemia with a distinct penumbra (at least 20%), measured by magnetic resonance perfusion imaging (PI) and diffusion-weighted imaging (DWI), in the territory of the middle cerebral artery, anterior cerebral artery, or posterior cerebral artery with a hemispheric distribution
5. Ability and willingness to provide informed consent and comply with study requirements and procedures

Exclusion Criteria:

1. Eligibility for acute thrombolytic (rtPA) treatment
2. Normal brain MRI
3. Transient ischemic attack or rapidly improving neurological symptoms
4. Previous disability
5. Hemorrhagic stroke on brain MRI (T2*/SWI)
6. Ongoing infection defined by clinical and laboratory signs: an evidence-based guideline will be followed to detect infectious complications (in short, physical and laboratory measures including WBC, ESR, hsCRP, PCT, fever, abnormal urine, chest X-ray or positive cultures)
7. Diagnosis of malignancy
8. Known sensitivity to any ingredients in the study drug or radiological contrast material
9. Participation in another clinical trial within the past 30 days
10. Stroke in the previous 3 months
11. Chronic liver, kidney or hematological disease
12. Contraindications to MRI -Brain aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or defibrillator, cochlear implant, ocular foreign body e.g. metal shavings, other implanted medical devices: (e.g. Swan Ganz catheter) insulin pump, metal shrapnel or bullet.
13. Diabetes
14. Hypertension
15. Females who are pregnant or breastfeeding

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Post-IVIG DWI/PI mismatch measurement | 3 days
  Decrease in the size of post IVIG necrotic area relative to baseline values and percent of penumbra saved, defined by neuroimaging as DWI/PI mismatch.

SECONDARY OUTCOMES:
Favorable clinical outcome | 90 days
  Favorable clinical outcome at Day 90, which requires fulfillment of all three of the following criteria: improvement in NIHSS of 8 points or more from baseline; modified Rankin scale (mRS) score of 0-2 points; and Barthel index (BI) of 75-100
Clinical outcome measure by NIHSS | 3 days
  Clinical outcome measured by change in NIHSS scores will be also examined on Day 3
Active complement fragment levels | 90 days
  Levels of active complement fragments, C3a, C5a, C5b-9 and C4d at Day 0 and post-IVIG and Day 90.
Adverse Events | 90 days
  Incidence in adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly C Walters, MD, Study Director — Inova Health Systems; Milan Basta, MD, Study Chair — BioVisions, Inc.; Jack Cochran, MD, Principal Investigator — Inova Health Systems
Locations (1):
- Inova Health Systems; Inova Fairfax Hospital, Falls Church, Virginia, United States

REFERENCES:
- [Background] D'Ambrosio AL, Pinsky DJ, Connolly ES. The role of the complement cascade in ischemia/reperfusion injury: implications for neuroprotection. Mol Med. 2001 Jun;7(6):367-82. PMID 11474130
- [Background] Ember JA, Hugli TE. Complement factors and their receptors. Immunopharmacology. 1997 Dec;38(1-2):3-15. doi: 10.1016/s0162-3109(97)00088-x. PMID 9476110
- [Background] de Boer JP, Wolbink GJ, Thijs LG, Baars JW, Wagstaff J, Hack CE. Interplay of complement and cytokines in the pathogenesis of septic shock. Immunopharmacology. 1992 Sep-Oct;24(2):135-48. doi: 10.1016/0162-3109(92)90019-9. PMID 1473964
- [Background] Szalai AJ, van Ginkel FW, Wang Y, McGhee JR, Volanakis JE. Complement-dependent acute-phase expression of C-reactive protein and serum amyloid P-component. J Immunol. 2000 Jul 15;165(2):1030-5. doi: 10.4049/jimmunol.165.2.1030. PMID 10878380
- [Background] Van Beek J, Bernaudin M, Petit E, Gasque P, Nouvelot A, MacKenzie ET, Fontaine M. Expression of receptors for complement anaphylatoxins C3a and C5a following permanent focal cerebral ischemia in the mouse. Exp Neurol. 2000 Jan;161(1):373-82. doi: 10.1006/exnr.1999.7273. PMID 10683302
- [Background] Lindsberg PJ, Ohman J, Lehto T, Karjalainen-Lindsberg ML, Paetau A, Wuorimaa T, Carpen O, Kaste M, Meri S. Complement activation in the central nervous system following blood-brain barrier damage in man. Ann Neurol. 1996 Oct;40(4):587-96. doi: 10.1002/ana.410400408. PMID 8871578
- [Background] Nishino H, Czurko A, Fukuda A, Hashitani T, Hida H, Karadi Z, Lenard L. Pathophysiological process after transient ischemia of the middle cerebral artery in the rat. Brain Res Bull. 1994;35(1):51-6. doi: 10.1016/0361-9230(94)90215-1. PMID 7953757
- [Background] Figueroa E, Gordon LE, Feldhoff PW, Lassiter HA. The administration of cobra venom factor reduces post-ischemic cerebral injury in adult and neonatal rats. Neurosci Lett. 2005 May 20-27;380(1-2):48-53. doi: 10.1016/j.neulet.2005.01.027. Epub 2005 Feb 2. PMID 15854749
- [Background] Arumugam TV, Tang SC, Lathia JD, Cheng A, Mughal MR, Chigurupati S, Magnus T, Chan SL, Jo DG, Ouyang X, Fairlie DP, Granger DN, Vortmeyer A, Basta M, Mattson MP. Intravenous immunoglobulin (IVIG) protects the brain against experimental stroke by preventing complement-mediated neuronal cell death. Proc Natl Acad Sci U S A. 2007 Aug 28;104(35):14104-9. doi: 10.1073/pnas.0700506104. Epub 2007 Aug 21. PMID 17715065
- [Background] Szeplaki G, Szegedi R, Hirschberg K, Gombos T, Varga L, Karadi I, Entz L, Szeplaki Z, Garred P, Prohaszka Z, Fust G. Strong complement activation after acute ischemic stroke is associated with unfavorable outcomes. Atherosclerosis. 2009 May;204(1):315-20. doi: 10.1016/j.atherosclerosis.2008.07.044. Epub 2008 Aug 14. PMID 18804761
- [Background] De Simoni MG, Rossi E, Storini C, Pizzimenti S, Echart C, Bergamaschini L. The powerful neuroprotective action of C1-inhibitor on brain ischemia-reperfusion injury does not require C1q. Am J Pathol. 2004 May;164(5):1857-63. doi: 10.1016/S0002-9440(10)63744-3. PMID 15111332
- [Background] De Simoni MG, Storini C, Barba M, Catapano L, Arabia AM, Rossi E, Bergamaschini L. Neuroprotection by complement (C1) inhibitor in mouse transient brain ischemia. J Cereb Blood Flow Metab. 2003 Feb;23(2):232-9. doi: 10.1097/01.WCB.0000046146.31247.A1. PMID 12571454
- [Background] Akita N, Nakase H, Kaido T, Kanemoto Y, Sakaki T. Protective effect of C1 esterase inhibitor on reperfusion injury in the rat middle cerebral artery occlusion model. Neurosurgery. 2003 Feb;52(2):395-400; discussion 400-1. doi: 10.1227/01.neu.0000043710.61233.b4. PMID 12535370
- [Background] Akita N, Nakase H, Kanemoto Y, Kaido T, Nishioka T, Sakaki T. [The effect of C 1 esterase inhibitor on ischemia: reperfusion injury in the rat brain]. No To Shinkei. 2001 Jul;53(7):641-4. Japanese. PMID 11517488
- [Background] Basta M, Fries LF, Frank MM. High doses of intravenous Ig inhibit in vitro uptake of C4 fragments onto sensitized erythrocytes. Blood. 1991 Jan 15;77(2):376-80. PMID 1985703
- [Background] Basta M, Langlois PF, Marques M, Frank MM, Fries LF. High-dose intravenous immunoglobulin modifies complement-mediated in vivo clearance. Blood. 1989 Jul;74(1):326-33. PMID 2752117
- [Background] Basta M, Kirshbom P, Frank MM, Fries LF. Mechanism of therapeutic effect of high-dose intravenous immunoglobulin. Attenuation of acute, complement-dependent immune damage in a guinea pig model. J Clin Invest. 1989 Dec;84(6):1974-81. doi: 10.1172/JCI114387. PMID 2687331
- [Background] Basta M. Modulation of complement-mediated immune damage by intravenous immune globulin. Clin Exp Immunol. 1996 May;104 Suppl 1:21-5. PMID 8625538
- [Background] Basta M, Van Goor F, Luccioli S, Billings EM, Vortmeyer AO, Baranyi L, Szebeni J, Alving CR, Carroll MC, Berkower I, Stojilkovic SS, Metcalfe DD. F(ab)'2-mediated neutralization of C3a and C5a anaphylatoxins: a novel effector function of immunoglobulins. Nat Med. 2003 Apr;9(4):431-8. doi: 10.1038/nm836. Epub 2003 Mar 3. PMID 12612546
- [Background] Basta M. Ambivalent effect of immunoglobulins on the complement system: activation versus inhibition. Mol Immunol. 2008 Oct;45(16):4073-9. doi: 10.1016/j.molimm.2008.07.012. Epub 2008 Aug 15. PMID 18706699
- [Background] Spycher M, Matozan K, Minnig K, Zehnder R, Miescher S, Hoefferer L, Rieben R. In vitro comparison of the complement-scavenging capacity of different intravenous immunoglobulin preparations. Vox Sang. 2009 Nov;97(4):348-54. doi: 10.1111/j.1423-0410.2009.01217.x. Epub 2009 Jul 27. PMID 19656348
- [Background] Al-Buhairi AR, Jan MM. Recombinant tissue plasminogen activator for acute ischemic stroke. Saudi Med J. 2002 Jan;23(1):13-9. PMID 11938357
- [Background] Clark WM, Wissman S, Albers GW, Jhamandas JH, Madden KP, Hamilton S. Recombinant tissue-type plasminogen activator (Alteplase) for ischemic stroke 3 to 5 hours after symptom onset. The ATLANTIS Study: a randomized controlled trial. Alteplase Thrombolysis for Acute Noninterventional Therapy in Ischemic Stroke. JAMA. 1999 Dec 1;282(21):2019-26. doi: 10.1001/jama.282.21.2019. PMID 10591384
- [Background] Bennett WR, Yawn DH, Migliore PJ, Young JB, Pratt CM, Raizner AE, Roberts R, Bolli R. Activation of the complement system by recombinant tissue plasminogen activator. J Am Coll Cardiol. 1987 Sep;10(3):627-32. doi: 10.1016/s0735-1097(87)80206-1. PMID 3114350
- [Background] Szeplaki G, Varga L, Laki J, Dosa E, Madsen HO, Prohaszka Z, Szabo A, Acsady G, Selmeci L, Garred P, Fust G, Entz L. Elevated complement C3 is associated with early restenosis after eversion carotid endarterectomy. Thromb Haemost. 2006 Oct;96(4):529-34. PMID 17003933
- [Background] Darabi K, Abdel-Wahab O, Dzik WH. Current usage of intravenous immune globulin and the rationale behind it: the Massachusetts General Hospital data and a review of the literature. Transfusion. 2006 May;46(5):741-53. doi: 10.1111/j.1537-2995.2006.00792.x. PMID 16686841
- [Background] Ahsan N, Palmer BF, Wheeler D, Greenlee RG Jr, Toto RD. Intravenous immunoglobulin-induced osmotic nephrosis. Arch Intern Med. 1994 Sep 12;154(17):1985-7. doi: 10.1001/archinte.154.17.1985. PMID 8074604
- [Background] Bednarik J, Kadanka Z. [Adverse effects of administration of intravenous human immunoglobulins]. Cas Lek Cesk. 1999 Nov 1;138(21):647-9. Czech. PMID 10746020
- [Background] Orbach H, Katz U, Sherer Y, Shoenfeld Y. Intravenous immunoglobulin: adverse effects and safe administration. Clin Rev Allergy Immunol. 2005 Dec;29(3):173-84. doi: 10.1385/CRIAI:29:3:173. PMID 16391392
- [Background] Al-Wahadneh AM, Khriesat IA, Kuda EH. Adverse reactions of intravenous immunoglobulin. Saudi Med J. 2000 Oct;21(10):953-6. PMID 11369961
- [Background] Katz U, Shoenfeld Y. Review: intravenous immunoglobulin therapy and thromboembolic complications. Lupus. 2005;14(10):802-8. doi: 10.1191/0961203303lu2168rr. PMID 16302674
- [Background] Reinhart WH, Berchtold PE. Effect of high-dose intravenous immunoglobulin therapy on blood rheology. Lancet. 1992 Mar 14;339(8794):662-4. doi: 10.1016/0140-6736(92)90806-e. PMID 1347348
- [Background] Fisher M. Characterizing the target of acute stroke therapy. Stroke. 1997 Apr;28(4):866-72. doi: 10.1161/01.str.28.4.866. PMID 9099209
- [Background] Lansberg MG, O'Brien MW, Tong DC, Moseley ME, Albers GW. Evolution of cerebral infarct volume assessed by diffusion-weighted magnetic resonance imaging. Arch Neurol. 2001 Apr;58(4):613-7. doi: 10.1001/archneur.58.4.613. PMID 11295992